CLINICAL TRIAL: NCT07364331
Title: Omega- 3 Fatty Acids, Neuroendocrine and Attention Deficit Hyperactivity Disorder With (OMNeADHD) A Double Blind Randomized Controlled Trial of High Dose Omega- 3 Fatty Acids in Children and Adolescents With ADHD With Omega- 3 Deficiency.
Brief Title: Omega-3 Fatty Acids, Neuroendocrine and Attention Deficit Hyperactivity Disorder (OMNeADHD)
Acronym: OMNeADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Pei-Chen Chang, Director of Child Psychiatry Division, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH110-REC3-203
Record Dates: First submitted 2024-04-25; First posted 2026-01-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: ADHD; Children; Adolescents
Keywords: omega-3; epa; dha; children; ADHD; adolescents
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: This is a 12 week study to investigate the effects of EPA, DHA and placebo in youth with ADHD
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- omega-3 fatty acids: EPA (Active Comparator): EPA
  Interventions: Dietary Supplement: Omega-3
- omega-3 fatty acids: DHA (Active Comparator): DHA
  Interventions: Dietary Supplement: Omega-3
- placebo (Placebo Comparator): olive oil
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 — EPA or DHA
  Arms: omega-3 fatty acids: DHA; omega-3 fatty acids: EPA
Dietary Supplement: Placebo — olive oil
  Arms: placebo

SUMMARY:
This is a 12 week randomized controlled study on the effects of omega-3 fatty acids in youth with attention deficit hyperactivity disorder (ADHD) with omega-3 deficiency.

DETAILED DESCRIPTION:
This is a 12 week randomized controlled study on the effects of omega-3 fatty acids (EPA or DHA) in youth with attention deficit hyperactivity disorder (ADHD) with omega-3 deficiency.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-5 diagnosis of ADHD
2. Did not have any changes of ADHD treatment (pharmacological/psychological) within 4 weeks of entering the trial.
3. SNAP-IV inattention subscale >=12, or hyperactivity subscale >=12, or inattention+ hyperactivity subscales >=24

Exclusion Criteria:

1. IQ<80
2. Allergic to omega-3
3. Physical disorders: thyroid function, cancer
4. Psychiatric comorbidity: SUD, psychotic disorders, bipolar disorder, major depressive disorder

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-04 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Clinical symptoms-attention and impulsivity symptom severity | week 0,1,2,4,8,12
  The Swanson, Nolan, and Pelham Rating Scale- 4th edition (SNAP-IV) is used to help assess symptoms of ADHD (Attention Deficit Hyperactivity Disorder) in children and adolescents. It consists of a series of questions that rate the severity of behaviors such as inattention, hyperactivity, and impulsivity, based on teacher and parent observations. The scale includes both parent and teacher versions, allowing for a comprehensive view of a child's behavior in different environments. The scoring system rates each behavior on a 4-point scale from 0 (never or rarely) to 3 (very often), and higher total scores indicate more significant ADHD symptoms. The results help clinicians in diagnosing ADHD and monitoring treatment progress.

SECONDARY OUTCOMES:
Measurement of cognitive function: attention and impulsivity | week 0,12
  The Continuous Performance Test (CPT) will be used to measure attention and impulse control of the subjects. During the test, individuals are presented with a series of stimuli and must respond to specific targets while ignoring distractions. It is commonly used to assess attention deficits and impulsivity, key symptoms in ADHD.
Concentration of Peripheral cortisol levels | week 0,12
  saliva and blood samples will be taken to assess peripheral cortisol levels. (micrograms/deciliter, μg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Chen Chang, PhD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No